CLINICAL TRIAL: NCT03431051
Title: The Impact of Workplace Food and Beverage Choices on Health and Wellness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Laura and John Arnold Foundation (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jamey Schmidt, Director, Clinical Research, California Pacific Medical Center Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Healthy Beverage Initiative
Record Dates: First submitted 2018-01-29; First posted 2018-02-13 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Health and Wellness
Keywords: Healthy Beverage Initiative, Sugar Sweetened Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Beverage Initiative (Active Comparator): A Healthy Beverage Initiative and health education will be implemented at two hospital campuses.
  Interventions: Other: Healthy Beverage Initiative
- Control Arm (No Intervention): No change in beverages or education at two hospital campuses.

INTERVENTIONS:
Other: Healthy Beverage Initiative — A Healthy Beverage Initiative will be instituted at two hospital campuses.
  Arms: Healthy Beverage Initiative

SUMMARY:
The study is designed to determine if instituting a Healthy Beverage Initiative (HBI) at hospitals influences health and wellness of employees over a 12 month period.

DETAILED DESCRIPTION:
To examine whether HBI is associated with decreased adiposity over a 12-month time period, in comparison to individuals identically assessed but not exposed to a HBI. Specifically, do those exposed to the HBI decrease in measures of adiposity, BMI, and sugar sweetened beverage (SSB) intake? Do they decrease more in those measures as compared to those not exposed to the HBI?

ELIGIBILITY:
Inclusion Criteria:

* The participant speaks and reads English.
* The participant consumes three or more sugar-sweetened beverages a week.
* The participant expects to be able to participate for all 3 visits (baseline, 6 months, and 12 months).

Exclusion Criteria:

The participant is planning an extended leave of absence and/or family medical leave of absence over the next 12 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal adiposity | About one year.
  Study participants at HBI campuses will show improvements (specifically, decreases) in indices of abdominal adiposity measured using waist circumference in centimeters.
Abdominal adiposity | About one year.
  Study participants at HBI campuses will show improvements (specifically, decreases) in indices of abdominal adiposity measured using sagittal abdominal diameter in centimeters.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | About one year.
  Study participants at HBI campuses will show improvements (specifically, decreases) in body mass index [BMI] measured using height in centimeters and weight in kilograms to be calculated into BMI in kg/m^2.
Sugar Sweetened Beverage Intake | About one year.
  Study participants at HBI campuses will show improvements (specifically, decreases) in SSB intake measured by the BEVQ (beverage food frequency questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Greg Tranah, PhD, Study Director — Sutter Health-California Pacific Medical Center Research Institute
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States